CLINICAL TRIAL: NCT03984734
Title: Randomized Trial Comparing Quality of Life and Nutritional Status Between Pylorus-preserving Pancreatoduodenectomy Versus Standard Pancreatoduodenectomy (QUANUPAD TRIAL)
Brief Title: Quality of Life and Nutritional Status After Two Surgical Techniques in Pancreatoduodenectomy
Acronym: QUANUPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, BUSQUETS, JULI, Staff surgeon Bellvitge Universitary Hospital, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QUANUPAD
Record Dates: First submitted 2019-03-25; First posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Delayed Gastric Emptying
Keywords: Delayed Gastric Emptying; Pylorus-preserving pancreatoduodenectomy
MeSH Terms: conditions — Gastroparesis | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients undergoing pancreatoduodenectomy with antrectomy
  Interventions: Procedure: Pancreatoduodenectomy with antrectomy
- Study group (Experimental): Patients undergoing pancreatoduodenectomy with pylorus-preserving pancreatoduodenectomy
  Interventions: Procedure: Pylorus-preserving pancreatoduodenectomy

INTERVENTIONS:
Procedure: Pancreatoduodenectomy with antrectomy
  Arms: Control group
Procedure: Pylorus-preserving pancreatoduodenectomy
  Arms: Study group

SUMMARY:
This was a randomized unblinded single-centre trial. The main hypothesis of the study was that pylorus-preserving pancreatoduodenectomy reduces the incidence of delayed gastric emptying . Patients undergoing pancreatoduodenectomy were randomized to undergo one of two types of surgical technique: pylorus-preserving pancreatoduodenectomy versus stardard pancreatoduodenectomy with antrectomy. The primary endpoint was the incidence and severity of delayed gastric emptying. Secondary endpoints were postoperative morbidity and mortality, length of hospital stay, and nutritional status and quality of life.

DETAILED DESCRIPTION:
This was a randomized unblinded single-centre trial without masked evaluation of the main outcome.The authors decided to compare pancreatoduodenectomy with antrectomy versus pancreatoduodenectomy with pyloric preservation. The primary aim of this randomized clinical trial was to determine whether pancreatoduodenectomy with pyloric preservation is associated with a lower incidence and severity of delayed gastric emptying. Secondary endpoints were postoperative complications, postoperative mortality and duration of hospital stay. Patients undergoing pancreatoduodenectomy were randomized to undergo one of two types of gastroenteric anastomosis for reconstruction. Analytical parameters such as C-reactive protein, prealbumin, and albumin; as well as anthropometric measures (mean) as preoperative arm circumference mean and tricipital skinfold mean were registered preoperatively, at 5th week, and at 6th mounth. Scintigraphic study had performed following a specific protocol for gastric emptying. At the end, quality of life was also analized with a quality of life questionnaire (QLPAN26) preoperativelly and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgical resection of the head of the pancreas at the authors' institution from August 2003 to August 2008. Adults of either sex aged over 18 years were included.

Exclusion Criteria:

* Associated resections of other organs, except for the portal or superior mesenteric vein
* Total pancreatectomy
* Previous gastrectomy or other gastric surgeries
* Neoadjuvant treatment
* Liver cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of DGE | within the first 90 days after surgery
  Nasogastric tube not removed before the 10th postoperative days or if liquids were not tolerated before the 14th postoperative day

SECONDARY OUTCOMES:
Postoperative morbidity | within the first 90 days after surgery
  Appearance of any complication during the hospital stay
Postoperative mortality | within the first 90 days after surgery
  Any death that happens during the hospital admission or within 90 days after surgery
Length of hospital stay | within the first 90 days after surgery
  Postoperative hospital stay after pancreatoduodenectomy

CONTACTS AND LOCATIONS:
Overall Officials: Juan Fabregat Prous, Dr., Principal Investigator — Hospital Universitari de Bellvitge

REFERENCES:
- [Derived] Busquets J, Martin S, Secanella L, Sorribas M, Cornella N, Altet J, Pelaez N, Bajen M, Carnaval T, Videla S, Fabregat J. Delayed gastric emptying after classical Whipple or pylorus-preserving pancreatoduodenectomy: a randomized clinical trial (QUANUPAD). Langenbecks Arch Surg. 2022 Sep;407(6):2247-2258. doi: 10.1007/s00423-022-02583-9. Epub 2022 Jul 4. PMID 35786739